CLINICAL TRIAL: NCT05952128
Title: A Single-center, Prospective, Single-arm Phase Ib/II Clinical Study on the Efficacy and Safety of Fluzoparib Combined With Dalpiciclib in the Treatment of Locally Advanced or Metastatic Sarcoma r
Brief Title: Phase Ib/II Study of Fluzoparib in Combination With Dalpiciclib in Patients With Locally Advanced or Metastatic Sarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jin Wang,MD, Chief Physician Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2023-085-01
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Sarcoma
Keywords: Fluzoparib; Dalpiciclib
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluzoparib+ Dalpiciclib (Experimental): Fluzoparib in combination with Dalpiciclib
  Interventions: Drug: Fluzoparib+ Dalpiciclib

INTERVENTIONS:
Drug: Fluzoparib+ Dalpiciclib — Drug Fluzoparib 100mg bid PO qd, administered continuously until disease progression, unacceptable toxicity or death. 28 days as a treatment cycle.
  Other names: SHR-3162
  Drug Dalpiciclib 100mg/125mg/150mg PO qd, administered only from day1 to day 21 every cycle until disease progression, unacceptable toxicity or death. 28 days as a treatment cycle.
  Other names: SHR-6390

SUMMARY:
This is a single-center, single-arm phase Ib / II clinical trial, which was included with two phase. The main purpose of the phase Ib part was to determine the dose-limiting toxicity ( DLT ), maximum tolerated dose ( MTD ), and recommended dose ( RP2D ) of Fluzoparib combined with Dalpiciclib in patients with locally advanced or metastatic sarcoma. The phase II part is mainly to observe the efficacy and safety of Fluzoparib combined with Dalpiciclib.

DETAILED DESCRIPTION:
The overall prognosis for patients with soft tissue sarcoma is not ideal, with a median survival rate of only about 20 months for patients diagnosed with metastasis. Soft tissue sarcomas (more than 50%) are deficient in HRR due to the presence of BRCA mutations in the tumor. When patients with BRCA1/2 gene mutation are treated with PARP inhibitors, a damage to DNA single strand breaks can be observed, and cannot be repaired promptly, resulting in tumor cell death. In addition, selective inhibition of CDK4/6 was found to inhibit the growth of sarcoma cells and induce their apoptosis. For example, inhibition of CDK4 decrease the proliferation of osteosarcoma cells and promote their apoptosis in vitro, and targeted CDK6 inhibition can inhibit the proliferation, invasion and migration of Ewing's sarcoma cells. Therefore, in this study, Dalpicicli, a CDK4/6 inhibitor, and Fluzoparib, a PARP inhibitor, were used in the treatment of advanced and metastatic soft tissue sarcoma, so as to explore the efficacy and safety of the combined regimen.

ELIGIBILITY:
Inclusion Criteria:1.Patients aged 12 to 75 years, male and female ; 2.Eastern Cooperative Oncology Group ( ECOG ) physical status score was 0-2 ; 3.Locally advanced or metastatic sarcomas ( including osteosarcoma, Ewing sarcoma, undifferentiated sarcoma, liposarcoma, leiomyosarcoma, fibrosarcoma and synovial sarcoma ) confirmed by histopathology, and at least one measurable lesion without local treatment ( according to RECIST v1.1, the long diameter of the measurable lesion mesured by spiral CT scan should be≥ 10 mm or the short diameter of the lymph node lesion should be ≥ 15 mm ) ; 4.Life expectancy≥ 12 weeks ; 5.The main organ function is basically normal and meets the program requirements :

a)Blood examination : (without blood transfusion within 14 days before screening, without using granulocyte colony stimulating factor [ G-CSF ], or other methods to correct bone marrow suppression within 7 days ) ,Blood indicators should meet: i.hemoglobin ≥ 90 g / L ; ii.neutrophil count ≥ 1.5 × 109 / L ; iii.Platelet count ≥ 75 × 109 / L ; b)b. Biochemical examination : ( no albumin transfusion within 14 days ) indicators should meet: i.albumin ≥ 29 g / L ; ii.Alanine aminotransferase ( ALT ) and aspartate aminotransferase ( AST ) ≤ 2.5 times the upper limit of normal ( ULN ) ; iii.total bilirubin ( TBIL ) ≤ 1.5 times ULN ; iv.Creatinine Cr ≤ 1.5 times ULN or Cr clearance > 50 mL / min; v.Urine protein < 2 +. If Urine protein ≥ 2 +, an 24 hours ( h ) urine protein quantification test should be taken, and 24h urine protein quantification < 1.0 g is allowed to include ) ; c)Coagulation function : activated partial thromboplastin time ( APTT ) and international normalized ratio ( INR ) ≤ 1.5 × ULN ( for those who regularly use anticoagulant therapy such as low molecular weight heparin or warfarin and INR meets the expected requirement are allowed to include ) ; d)Thyroid stimulating hormone ( TSH ) ≤ ULN ; If not, T3 and T4 levels should be examined, and only with normal T3 and T4 level is allowed to include.

e)Echocardiography : left ventricular ejection fraction ( LVEF ) ≥ 60 %. 6.Non-surgical sterilization or women of childbearing age who are required to use a medically approved contraceptive (such as an intrauterine device, contraceptive pill or condom) during the study treatment period and for 6 months after the study treatment period ends; Female patients of childbearing age who were not surgically sterilized must have a negative serum or urine HCG test within 7 days prior to study enrollment; And must be non-lactation period; For male patients with a partner of a woman of childbearing age, effective contraceptive methods should be used during the trial period and within 6 months after the last Fluzoparib or Dalpiciclib administration.

Understand the research procedures and methods, volunteer to participate in the experiment, and sign the informed consent. And fully understand the trial content, process and possible adverse reactions.

-

Exclusion Criteria:1.Plan to receive any other antitumor therapy during this trial; 2.Within 4 weeks of the first administration of the drug in this study, the patient has received radiotherapy for sarcoma, or received compound names such as Fluzoparib, Dalpiciclib, drug administration or cell therapy in other clinical trials; 3.Imaging diagnosis showed the presence of tumor lesions in the brain; 4.Active malignancies other than sarcoma within 5 years or at the same time. Cured localized tumors, such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder carcinoma, prostate carcinoma in situ, cervical carcinoma in situ, breast carcinoma in situ, etc., could be included in the group.

5.Patients with clinical symptoms of ascites requiring puncture or drainage, or patients who have received ascites drainage within the past 3 months, except those who only show a small amount of ascites without clinical symptoms on imaging; Uncontrolled or medium or above pleural effusion and pericardial effusion; There is evidence of abdominal gas accumulation that cannot be explained by puncture or recent surgical procedures 6.Have a history of epilepsy, or a history of seizures within 12 months prior to the first administration of the study drug (including a history of transient ischemic attack, cerebral stroke (except imaging only found ischemic focus but no corresponding clinical history), brain trauma with disturbance of consciousness requiring hospitalization); 7.Previous treatment with PARP or CDK4/6 inhibitors, including but not limited to Fluzoparib and Dalpiciclib; 8.Allergic constitution, including severe drug allergy or drug allergic reaction history; Known allergies or intolerances to Fluzoparib, Dalpiciclib or their excipients; 9.Severe infections (CTC AE ≥grade 2), such as severe pneumonia, bacteremia, and infection complications requiring hospitalization, occurred within 4 weeks prior to the first use of the study drug; Baseline chest imaging suggests active pulmonary inflammation, signs and symptoms of infection within 2 weeks prior to the first use of the study drug, or the need for oral or intravenous use of the drug · Antibiotic therapy (excluding the use of prophylactic antibiotics); 10.Drugs that may affect P-gp should not be discontinued during the study； 11.Had use of a potent/moderate-acting drug that inhibits or induces the liver drug metabolizing enzyme CYP3A4 14 days prior to initial administration； 12.Inability to swallow, chronic diarrhea, intestinal obstruction, or other factors affecting drug administration and absorption; 13.A history of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML), or other malignancies (other than carcinoma in situ with complete response and malignancies determined by the investigator to be slow in progression) within 5 years prior to the initial administration of the study; 14.Combined with other viral infection (anti-HCV, anti-HIV positive, HBsAg positive) or syphilis infection; 15.A history of immunodeficiency (including HIV test positive, other acquired or congenital immunodeficiency diseases) or a history of organ transplantation; 16.A known history of psychotropic drug abuse, alcoholism and drug use; A concomitant disease (such as poorly controlled hypertension, severe diabetes, thyroid disease, and psychosis) or any other condition that, in the investigator's judgment, seriously endangers the patient's safety or affects the patient's ability to complete the study.

-

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase II dose (RP2D) | from 4 weeks to 20 weeks after the first dose of Fluzoparib and Dalpiciclib combination therapy
  Determination of Recommended Phase II dose (RP2D) of Escalating Dose of Fluzoparib with Dalpiciclib.
dose limiting toxicity (DLT). | from 4 weeks to 20 weeks after the first dose of Fluzoparib and Dalpiciclib combination therapy
  Observe the incidence of dose limiting toxicity (DLT).
maximize toxicity dose(MTD) | from 4 weeks to 20 weeks after the first dose of Fluzoparib and Dalpiciclib combination therapy
  Determination of maximize toxicity dose(MTD)
Objective Response Rate(ORR) as Assessed by the Investigator according to RECIST v1.1 | up to approximately 2 Years
  Objective Response Rate(CR+PR), defined as best overall response (complete or partial response) across all assessment time points, determined using RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Disease control rate(DCR) | Up to approximately 2 Years
  Disease control rate(DCR) is defined DCR=CR+PR+SD/CR+PR+SD+PD, which reflects the ratio of patients whose tumors shrank or remained stable for a certain period of time.
Duration of remisson(DoR) | Up to approximately 2 Years
  Duration of remisson(DoR) is defined as the time interval from the beginning of the response ( when CR or PR is first determined ) to progression or death ( whichever occurs first ).
Progression free surviral(PFS) | Up to approximately 2 Years
  Progression Free Survival is defined as from the date of first administration to the date of disease progression or death, no matter which is earlier.
Overall survial(OS) | Up to approximately 2 Years
  Overall survial(OS) is defined as from the date of first administration to the date of death.
Incidence of Adverse Events [safety and tolerability] | From the first administration to 30 days after the last administration
  Adverse events defined according to Common Terminology for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: wangjinr@sysucc.org.cn Wang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer Center of Sun-Yat Sen University (CCSYSU), Guangzhou, Guangdong, China